CLINICAL TRIAL: NCT07406620
Title: Entropy-Based Assessment of Physiological Signals in Obstructive Sleep Apnoea Patients Pre and Post Continuous Positive Airway Pressure Therapy: A Secondary Analysis of 3DPiPPIn Trial Data
Brief Title: Entropy-based Physiological Signal Analysis in Patients With Obstructive Sleep Apnoea
Acronym: EPPOSA
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Ime Umoabasi, MRes Clinical Research Student, King's College London
Other Study IDs: 366646
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnoea (OSA)
Keywords: Obstructive Sleep Apnoea; OSA; Continous Positive Airway Pressure; CPAP; Entropy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3DPiPPIn Trial Participants: Participants were originally recruited to the 3DPiPPIn trial from the Sleep and Ventilation Service at Royal Free London NHS Foundation Trust. The cohort for this secondary analysis comprises adults with sleep-disordered breathing and an Apnoea-Hypopnoea Index (AHI) >15 events/hour who required but had never received PAP therapy, drawn from the trial participants who provided consent for their data to be used in future research.
  Interventions: Device: Continuous Positive Airway Pressure Therapy

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Therapy — The intervention of interest within this secondary analysis study is Continuous Positive Airway Pressure (CPAP) Therapy, a device-based treatment used to maintain airway patency in patients with sleep-disordered breathing. As a retrospective study, participant exposure to CPAP occured exclusively within the original 3DPiPPIn trial.
  Other Names: CPAP; CPAP Therapy; PAP; PAP Therapy; Positive Airway Pressure Therapy

SUMMARY:
This observational study is being undertaken as a part of a Master of Research (MRes) in Clinical Research programme.

Its goal is to learn about how continuous positive airway pressure (CPAP) therapy changes the complexity of body signals in adults with obstructive sleep apnoea (OSA). The main question it aims to answer is:

- How does the complexity of physiological signals (specifically oxygen saturation, heart rate variability, and airflow) change in adults with OSA from before to after three and six months of CPAP treatment?

It will use data from individuals who took part in an earlier trial, called 3DPiPPIn, which tested the use of 3D-printed, customised masks CPAP masks through sleep studies.

DETAILED DESCRIPTION:
The purpose of this MRes student study is primarily to examine how the entropy, or complexity as measured by entropy, of physiological signals changes in patients with obstructive sleep apnoea (OSA) in response to continuous positive airway pressure (CPAP) therapy.

It is a secondary analysis of data from 3DPiPPIn, a randomised control trial investigating the feasibility of using 3D-printing to develop customised masks for patients receiving positive airway pressure (PAP) therapy.

The hypothesis for this study is that entropy-based measures derived from physiological signals will exhibit changes following CPAP therapy, when compared to pre-therapy measures, reflecting the modulation and restoration of physiological systems that were previously disrupted by OSA.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the 3DPiPPIn trial
* Completion of the 3DPiPPIn trial to its primary endpoint of six months
* Availability of physiological signal data at baseline, three months, and six months
* Provision of informed consent permitting the use of their data in future research

Exclusion Criteria:

* Non-completion of the 3DPiPPIn trial to its primary endpoint of six months
* Missing physiological signal data at baseline, three months, or six months
* No consent for the use of their data in future research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAP-naive adults with obstructive sleep apnea (OSA), identified from the Sleep and Ventilation Service at Royal Free London NHS Foundation Trust, who participated in the 3DPiPPIn randomised controlled trial.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in oxygen saturation entropy from pre to six months post CPAP therapy | From baseline to six months post-initiation of CPAP therapy
Change in heart rate variability entropy from pre to six months post CPAP therapy | From baseline to six months post-initiation of CPAP therapy
Change in airflow entropy from pre to six months post CPAP therapy | From baseline to six months post-initiation of CPAP therapy

SECONDARY OUTCOMES:
Change in oxygen saturation entropy from pre to three months post CPAP therapy | From baseline to three months post-initiation of CPAP therapy
Change in heart rate variability entropy from pre to three months post CPAP therapy | From baseline to three months post-initiation of CPAP therapy
Change in airflow entropy from pre to three months post CPAP therapy | From baseline to three months post-initiation of CPAP therapy
Relationship between residual Apnoea-Hypopnoea Index and oxygen saturation entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Apnoea-Hypopnoea Index (AHI) is the total number of apnoea and hypopnoea events per hour of sleep. The minimum value is 0 events/hour, and there is no fixed maximum value. Higher scores indicate more severe sleep-disordered breathing (worse outcome).
Relationship between residual Apnoea-Hypopnoea Index and heart rate variability entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Apnoea-Hypopnoea Index (AHI) is the total number of apnoea and hypopnoea events per hour of sleep. The minimum value is 0 events/hour, and there is no fixed maximum value. Higher scores indicate more severe sleep-disordered breathing (worse outcome).
Relationship between residual Apnoea-Hypopnoea Index and airflow entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Apnoea-Hypopnoea Index (AHI) is the total number of apnoea and hypopnoea events per hour of sleep. The minimum value is 0 events/hour, and there is no fixed maximum value. Higher scores indicate more severe sleep-disordered breathing (worse outcome).
Relationship between Epworth Sleepiness Scale scores and oxygen saturation entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire that measures daytime sleepiness. Scores range from 0 to 24, with higher scores indicating greater daytime sleepiness (worse outcome).
Relationship between Epworth Sleepiness Scale scores and heart rate variability entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire that measures daytime sleepiness. Scores range from 0 to 24, with higher scores indicating greater daytime sleepiness (worse outcome).
Relationship between Epworth Sleepiness Scale scores and airflow entropy | From baseline to three and/or six months post-initiation of CPAP therapy
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire that measures daytime sleepiness. Scores range from 0 to 24, with higher scores indicating greater daytime sleepiness (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Izaak Neri, Study Director — King's College London; Stephanie K Mansell, Study Director — Royal Free London NHS Foundation Trust, University College London
Locations (2):
- United Kingdom (2):
  - Royal Free Hospital, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No
The data used in this secondary analysis include potentially re-identifiable patient information. In line with the open access approach of the study's parent trial, 3DPiPPIn, individual participant data will not be shared to protect participant confidentiality.

REFERENCES:
- [Background] Shah AJ. The use of wearable technology in chronic respiratory disease. Doctor of Philosophy (PhD), University College London; 2025. Available from: https://discovery.ucl.ac.uk/id/eprint/10212804
- [Background] Mansell SK, Mandal S, Ridout D, Olsen O, Gowing F, Kilbride C, Hilton ST, Main E, Schievano S. Clinical impact of customised positive airway pressure (PAP) therapy interfaces versus usual care in the treatment of patients with sleep-disordered breathing (3DPiPPIn): a randomised controlled trial protocol. BMJ Open. 2024 Nov 14;14(11):e087234. doi: 10.1136/bmjopen-2024-087234. PMID 39542493
- [Background] Mansell SK, Olsen O, Gowing F, Muwaffak Z, Kilbride C, Hilton S, Main E, Schievano S, Mandal S. 3DPiPPIN: 3D printing of positive airway pressure (PAP) therapy interfaces: a single site feasibility study. J Med Eng Technol. 2025 Oct;49(7):293-303. doi: 10.1080/03091902.2025.2532648. Epub 2025 Jul 29. PMID 40728908
- [Background] Mansell S, Olsen O, Smith L, Augustt S, Kilbride C, Ridout D, Hilton S, Main E, Schievano S, Mandal S. 3D Printing Positive Pressure Interfaces (3DPiPPIn): Results From a Two-Phase Feasibility Trial [Abstract]. Am J Respir Crit Care Med 2025;211:A6945. doi: 10.1164/ajrccm.2025.211.Abstracts.A6945